CLINICAL TRIAL: NCT03081702
Title: A Phase I/II Trial Investigating the Tolerability, Toxicity and Efficacy of Hydroxychloroquine and Itraconazole in Patients With Advanced Platinum-resistant Epithelial Ovarian Cancer (EOC) (HYDRA-1 Study)
Brief Title: A Study of the Safety, Tolerability and Effectiveness of Hydroxychloroquine and Itraconazole in Platinum-resistant Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYDRA-1
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Platinum-resistant Epithelial Ovarian Cancer
MeSH Terms: interventions — Hydroxychloroquine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxychloroquine and Itraconazole (Experimental): Hydroxychloroquine, orally (by mouth), at a dose of 100 mg, 200 mg, 400 mg, or 600 mg, twice a day, every day.
  Itraconazole, orally (by mouth) at 300 mg, twice a day, every day.
  Interventions: Drug: Hydroxychloroquine; Drug: Itraconazole

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine is approved/used for the treatment of rheumatoid arthritis, and discoid and systemic lupus erythematosus, as well as suppressive treatment and treatment of acute attacks of malaria.
Drug: Itraconazole — Itraconazole is approved and used for the treatment of certain systemic fungal infections.

SUMMARY:
This is a phase I/II study to find the highest dose of hydroxychloroquine that can be given safely with itraconazole in patients with advanced platinum-resistant epithelial ovarian cancer. The study will also determine the safety, tolerability, and initially determine whether the combination is useful in the treatment of patients with advanced platinum-resistant epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Histologically or cytologically confirmed epithelial ovarian cancer.
* Platinum-resistant or refractory disease defined as a radiological or clinical progression less than six months after having finished platinum-based chemotherapy.
* ECOG performance status equal to or less than 1.
* Have clinically or radiographically documented measurable disease.
* All systemic therapy must have been completed 4 weeks or greater prior to enrollment with radiologic evidence of radiological disease progression.
* Life expectancy should be more than 3 months.
* Receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible.
* Acceptable laboratory requirements within 7 days prior to enrollment
* Treated and asymptomatic brain metastases are eligible. Patients that received palliative radiation (for brain metastases) are eligible if they have been asymptomatic for at least 2 weeks with use of maintenance steroid therapy, and last received radiation at least 4 weeks prior to start of therapy.
* Have the ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Have not recovered (grade 1 or less) from adverse events related to previous treatments are excluded with the exception of alopecia and lymphopenia. Peripheral sensory neuropathy must be at grade 2 or less.
* Have any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site or any other cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to itraconazole or hydroxychloroquine.
* Known G6PD deficiency due to the risk of hemolytic anemia with the use of hydroxychloroquine.
* Known retinopathy due to the risk of worsening retinopathy with hydroxychloroquine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic or asymptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Chronic Hepatitis B or hepatitis C infections should be excluded because of potential effects on hepatic function and/ or drug interactions.
* Human Immunodeficiency Virus (HIV) infection.
* Already have a clinical indication for treatment with itraconazole (e.g. chronic candidiasis or other fungal infection) or hydroxychloroquine (e.g. lupus).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of hydroxychloroquine | 5 years
  Highest dose of hydroxychloroquine that is safe and tolerable that can be given in combination with itraconazole.

SECONDARY OUTCOMES:
Median progression-free survival | 5 years
  Median duration of time from start of treatment to time of progression or death.
Overall response rate | 5 years
  Proportion of patients achieving complete response or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marastoni S, Madariaga A, Pesic A, Nair SN, Li ZJ, Shalev Z, Ketela T, Colombo I, Mandilaras V, Cabanero M, Bruce JP, Li X, Garg S, Wang L, Chen EX, Gill S, Dhani NC, Zhang W, Pintilie M, Bowering V, Koritzinsky M, Rottapel R, Wouters BG, Oza AM, Joshua AM, Lheureux S. Repurposing Itraconazole and Hydroxychloroquine to Target Lysosomal Homeostasis in Epithelial Ovarian Cancer. Cancer Res Commun. 2022 May 4;2(5):293-306. doi: 10.1158/2767-9764.CRC-22-0037. eCollection 2022 May. PMID 36875717